CLINICAL TRIAL: NCT03733522
Title: Does the Isolation of the Operative Field Influence the Survival Rate of Bulkfill Composite Restorations in Primary Teeth
Brief Title: Isolation of the Operative Field Influences the Survival Rate of Composite Restorations
Acronym: IsolationC3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniela Prócida Raggio, Associated Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IsolationFOUSP
Record Dates: First submitted 2018-10-10; First posted 2018-11-07 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the evaluator of the restorations will be blind to the type of treatment (absolute or relative isolation). As the procedures are different, it will not be possible to blind operators and patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rubber dam isolation (Active Comparator): Absolute isolation
  * local anesthesia
  * use of dental clamp and rubber dam
  * restoration using Universal Adhesive in a self etch mode (Single Bond Universal - 3M ESPE) and bulkfill composite resin (Filtek Bulkfill - 3M ESPE)
  Interventions: Procedure: Relative isolation
- Relative isolation (Experimental): Relative isolation
  * no local anesthesia
  * use of cotton roll and saliva ejector
  * restoration using Universal Adhesive in a self etch mode (Single Bond Universal - 3M ESPE) and bulkfill composite resin (Filtek Bulkfill - 3M ESPE)
  Interventions: Procedure: Rubber dam isolation

INTERVENTIONS:
Procedure: Rubber dam isolation — Local anesthesia, use of dental clamp and rubber dam, followed by restoration using universal adhesive system and bulkfill composite restoration
  Arms: Relative isolation
Procedure: Relative isolation — No local anesthesia, use of cotton rollers and saliva ejector, followed by restoration using universal adhesive system and bulkfill composite restoration
  Arms: Rubber dam isolation

SUMMARY:
The aim of this study was to evaluate the survival of direct composite resin restorations in primary molars using different methods of isolation of the operative field: absolute isolation (local anesthesia, use of dental clamp and rubber dam) and relative isolation (cotton rollers and saliva ejector) by a randomized clinical trial. All composite restorations will be performed on children aged 4 to 10 years who present at least one dentin caries lesion or restoration needing replacement, without pulp involvement in a primary tooth. The treatments will be performed in the dental clinic of the University of São Paulo (FOUSP) by trained operators. The teeth will be randomized between the groups: Absolute Isolation (AI) and Relative Isolation (IR) and restored with composite resin (Scotchbond Universal Adhesive adhesive system and Filtek BulkFill composite resin - 3M ESPE) stratified by surface (single or multi surface). Restoration evaluation will be performed after 6, 12, 18, and 24 months by a blind, trained and calibrated examiner. As a primary outcome, the survival of the restorations will be evaluated. The secondary outcomes involve the procedure time (in minutes), professional and material cost (in Brazilian reais), as well as the cost-effectiveness of the restorations and the discomfort reported by the patient (measured using the Wong-Baker scale). The Kaplan-Meier survival analysis and log-rank test will be applied to the survival of the restoration. All variables will be modeled and compared with a Cox regression model of shared fragility. The discomfort reported by the patient will be analyzed by Ordinal Logistic Regression (α = 5%).

DETAILED DESCRIPTION:
Objective:

The aim of this study is to evaluate the survival of direct composite resin restorations in primary molars using different methods for isolation of the operative field: absolute isolation (local anesthesia, use of dental clamp and rubber dam) and relative isolation (cotton rollers and saliva ejector) by a randomized clinical trial.

Materials and Methods:

All composite restorations will be performed on children aged 4 to 10 years who present at least one dentin caries lesion or restoration needing replacement, without pulp involvement in a primary tooth. The treatments will be performed in the dental clinic of the University of São Paulo (FOUSP) by trained operators. The teeth will be randomized between the groups: Absolute Isolation (AI) and Relative Isolation (IR) and restored with composite resin (Scotchbond Universal Adhesive adhesive system and Filtek BulkFill composite resin - 3M ESPE) stratified by surface (single or multi surface).

Restoration evaluation will be performed after 6, 12, 18, and 24 months by a blind, trained and calibrated examiner.

As a primary outcome, the survival of the restorations will be evaluated. The secondary outcomes involve the procedure time (in minutes), professional and material cost (in Brazilian reais), as well as the cost-effectiveness of the restorations and the discomfort reported by the patient (measured using the Wong-Baker scale).

The Kaplan-Meier survival analysis and log-rank test will be applied to the survival of the restoration. All variables will be modeled and compared with a Cox regression model of shared fragility. The discomfort reported by the patient will be analyzed by Ordinal Logistic Regression (α = 5%).

ELIGIBILITY:
Inclusion Criteria:

* who have sought treatment in the University;
* between 4 and 10 years of age;
* with at least one dentin caries lesion without pulp involvement (ICCMS C score);
* need for restoration replacement diagnosed by FDI criteria or CARS criteria;
* absence of pulp involvement diagnosed by interproximal radiography (presence of dentin layer between the caries lesion and the pulp chamber).

Exclusion Criteria:

* children whose parents did not agree to participate in the study:
* children who did not agree to participate or had behavioral problems during the initial consultations.
* signs or symptoms of pulp pathology: spontaneous pain, pulp exposure, abscess or fistula near the tooth to be included, mobility or presence of communication between the caries lesion and the pulp (evaluated by interproximal digital radiography of the diagnosis).

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Survival of the restorations | Every 6 months up to 24 months
  The restorations will be evaluated according to the Roeleveld et al., 2006 criteria.
  Roeleveld et al. codes success (0-10) or failure (11-50).

SECONDARY OUTCOMES:
Child self-reported discomfort (0-5) | Immediately after treatment (in the same appointment)
  Wong-Baker Facial scale (Wong; Baker, 1998) from 0 to 5. The higher the score, higher the child self-reported discomfort.
Time spent during treatment (in minutes) | Immediately after treatment (in the same appointment)
  The total time spent in each restorative session will be recorded in minutes.
Procedure cost (in brazilian reais - R$) | Immediately after treatment (in the same appointment)
  Direct costs - all materials used in each procedure will be recorded. The average price of three different places in Brazilian market will be used (in Brazilian Reais).
Incremental Cost (in brazilian reais) | Every 12 months up to 24 months
  For the calculation of the final cost (Brazilian reais) of the treatment of each tooth will be used the result of the sum of the initial cost of the restorative procedure with the cost of repairs when necessary (incremental cost).

CONTACTS AND LOCATIONS:
Overall Officials: Daniela P Raggio, PhD, Study Director — University of Sao Paulo; Isabel C Olegário, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Background] Chisini LA, Collares K, Cademartori MG, de Oliveira LJC, Conde MCM, Demarco FF, Correa MB. Restorations in primary teeth: a systematic review on survival and reasons for failures. Int J Paediatr Dent. 2018 Mar;28(2):123-139. doi: 10.1111/ipd.12346. Epub 2018 Jan 10. PMID 29322626
- [Result] Roeleveld AC, van Amerongen WE, Mandari GJ. Influence of residual caries and cervical gaps on the survival rate of Class II glass ionomer restorations. Eur Arch Paediatr Dent. 2006 Jun;7(2):85-91. doi: 10.1007/BF03320820. PMID 17140533